CLINICAL TRIAL: NCT02334137
Title: Providing Diabetes Services in the Lions Eye Clinic: a Pilot Project to Assess the Impact of Diabetes Education During Ophthalmology Visits
Brief Title: A Pilot Project to Assess the Impact of Diabetes Education During Ophthalmology Visits
Acronym: LionsDMed
Status: Completed | Type: Observational
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Pacific Vision Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Diabetes Ed at Lions Eye
Record Dates: First submitted 2014-12-31; First posted 2015-01-08 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Complications; Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Complications; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- iPad app: This group will have unlimited access to educational iPad app while waiting for ophthalmology visits.
  Interventions: Behavioral: iPad app
- Educator sessions: This group will have unlimited access to educational iPad app AND at least one appointment with a certified diabetes educator or registered dietitian while waiting for ophthalmology visits.
  Interventions: Behavioral: iPad app; Behavioral: Educator sessions
- Educator sessions + retinal photos: This group will have same access as "iPad app + education sessions" and in addition will be able to briefly review their own retinal photos (compared to normal retina) with a resident ophthalmologist during timeline of pilot program.
  Interventions: Behavioral: iPad app; Behavioral: Educator sessions; Behavioral: Retinal photos

INTERVENTIONS:
Behavioral: iPad app — Provided by the Patient Education Institute, the "X-plain" iPad app includes modules on healthy eating for diabetics, eye complications, foot care, and others.
Behavioral: Educator sessions — A certified diabetes educator and/or registered dietitian will meet with patients for 30-60 minutes prior to their ophthalmology visits, when scheduling permits.
  Groups: Educator sessions; Educator sessions + retinal photos
Behavioral: Retinal photos — A resident ophthalmologist will spend approximately 5 minutes showing patient their own retinal photos, compared to a normal retina, and explaining the pathology present (if applicable).
  Groups: Educator sessions + retinal photos

SUMMARY:
The overarching purpose of this project is to provide diabetes education to the diverse patient population at the Lions Eye Clinic, a resident-run ophthalmology practice at California Pacific Medical Center. Because of high clinic volume in a teaching environment, our patients often experience long wait times. The goal of this program is to utilize this wait time for diabetes education, a much-needed corollary to the eye care that patients receive at our clinic.

This pilot project will investigate the impact of a program like this in our patient population. Specifically, the investigators are investigating whether diabetes education delivered in an ophthalmology setting enhances patient understanding of diabetes (via knowledge surveys) and/or leads to improved blood glucose control (via hemoglobin A1c). This is a 6-month study that runs through April 2015, and looks at the impact of an interactive diabetes education iPad app +/- in-person sessions with a diabetes educator. A subset of patients who meet with a diabetes educator will also be shown their own retinal images (compared to a normal retina).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes (as defined by evident systemic findings OR recent hemoglobin A1c OR patient report, as specific blood sugar data and knowledge of particular medications are often limited in this population)
* Age 18-75
* Able and willing to provide informed consent
* Speak English, Spanish, or any other language for which a translator is present

Exclusion Criteria:

* Advanced visual acuity loss in both eyes which prevents adequate use of educational tools
* Pregnant women, elderly patients (>75 years old), children and adolescents (17 or younger)
* Non-English/Spanish speakers for whom a translator is not present

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proposed subjects are diabetic patients already approved to be seen in the Lions Eye Clinic, specifically for dilated eye exam by a retinal specialist. This is a high-risk population with advanced disease and often with limited preexisting knowledge about diabetes, thus providing the motivation for these educational interventions.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Patient Knowledge about Diabetes at 3 months (via multiple-choice surveys) | Participants will be re-surveyed at their next follow-up eye appointment, an expected average of 3 months post-intervention
  Objective assessment of patient knowledge about diabetes using 13 multiple-choice questions

SECONDARY OUTCOMES:
Change from Baseline Hemoglobin A1c at 3 months | Participants will have repeat lab drawn at their next follow-up eye appointment, an expected average of 3 months post-intervention
  Provides estimate of patient's average blood sugar over past three months
Patient Satisfaction / Motivation / Subjective Improvement in Knowledge (brief surveys) | 1 day
  Brief 3-4 question surveys to assess patient satisfaction with services offered, motivation to manage their disease process, and subjective improvement in knowledge after using educational services
Change from Baseline in Patient Knowledge about Diabetes Immediately after using Educational Services (via multiple-choice surveys) | 1 day
  Objective assessment of patient knowledge about diabetes using 13 multiple-choice questions

CONTACTS AND LOCATIONS:
Overall Officials: Samuel J Reiter, MD, Study Director — Resident Ophthalmologist, CPMC; Taliva Martin, MD, Principal Investigator — CPMC Ophthalmologist, Residency Program Director